CLINICAL TRIAL: NCT06719479
Title: A Phase II/III Clinical Trial to Evaluate the Effect of IAE0972 Combined with Chemotherapy Selected by Doctors for Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma/Nasopharyngeal Carcinoma.
Brief Title: A Clinical Trial to Evaluate Effect of IAE0972 Combined with Chemotherapy for R/M HNSCC or NPC(Note: It is Currently Phase II.).
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAE0972-201
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: NPC; HNSCC; Recurrence; Metastasis
Keywords: NPC; HNSCC; Recurrence; Metastasis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 (Experimental): In Phase II，the patients will receive the combined treatment of IAE0972（7.5 mg/kg、10 mg/kg、15 mg/kg、20 mg/kg）+ Methotrexate（Chemotherapy chosen by doctors）. Every 21 days is defined as a treatment cycle.
  Interventions: Biological: IAE0972+ Methotrexate
- Cohort 2 (Experimental): In Phase II，the patients will receive the combined treatment of IAE0972（7.5 mg/kg、10 mg/kg、15 mg/kg、20 mg/kg）+ Docetaxel（Chemotherapy chosen by doctors）. Every 21 days is defined as a treatment cycle.
  Interventions: Biological: IAE0972+Docetaxel
- Cohort 3 (Experimental): In Phase II，the patients will receive the combined treatment of IAE0972（7.5 mg/kg、10 mg/kg、15 mg/kg、20 mg/kg）+ Gemcitabine（Chemotherapy chosen by doctors）. Every 21 days is defined as a treatment cycle.
  Interventions: Biological: IAE0972+Gemcitabine
- Cohort 4 (Experimental): In Phase II，the patients will receive the combined treatment of IAE0972（7.5 mg/kg、10 mg/kg、15 mg/kg、20 mg/kg）+ Taxanes （Chemotherapy chosen by doctors）. Every 21 days is defined as a treatment cycle.
  Interventions: Biological: IAE0972+Taxanes
- Cohort 5 (Experimental): In Phase II，the patients will receive the combined treatment of IAE0972（7.5 mg/kg、10 mg/kg、15 mg/kg、20 mg/kg）+ Capecitabine（Chemotherapy chosen by doctors）. Every 21 days is defined as a treatment cycle.
  Interventions: Biological: IAE0972+Capecitabine

INTERVENTIONS:
Biological: IAE0972+ Methotrexate — IAE0972: every 21 days is defined as a treatment cycle, and IAE0972 is infused intravenously on the 1d, 8d and 15d of each cycle. The first infusion time is about 120 min (which can be adjusted according to the actual situation); If the subjects are well tolerated when they receive the study drug for the first time (according to CTCAE 5.0, the infusion-related reaction is ≤ grade 1), the follow-up infusion time can be 60~90 min (which can be adjusted according to the actual situation).Methotrexate is used according to the instructions.
  Arms: Cohort 1
Biological: IAE0972+Docetaxel — IAE0972: every 21 days is defined as a treatment cycle, and IAE0972 is infused intravenously on the 1d, 8d and 15d of each cycle. The first infusion time is about 120 min (which can be adjusted according to the actual situation); If the subjects are well tolerated when they receive the study drug for the first time (according to CTCAE 5.0, the infusion-related reaction is ≤ grade 1), the follow-up infusion time can be 60~90 min (which can be adjusted according to the actual situation).Docetaxel is used according to the instructions.
  Arms: Cohort 2
Biological: IAE0972+Gemcitabine — IAE0972: every 21 days is defined as a treatment cycle, and IAE0972 is infused intravenously on the 1d, 8d and 15d of each cycle. The first infusion time is about 120 min (which can be adjusted according to the actual situation); If the subjects are well tolerated when they receive the study drug for the first time (according to CTCAE 5.0, the infusion-related reaction is ≤ grade 1), the follow-up infusion time can be 60~90 min (which can be adjusted according to the actual situation).Gemcitabine is used according to the instructions.
  Arms: Cohort 3
Biological: IAE0972+Taxanes — IAE0972: every 21 days is defined as a treatment cycle, and IAE0972 is infused intravenously on the 1d, 8d and 15d of each cycle. The first infusion time is about 120 min (which can be adjusted according to the actual situation); If the subjects are well tolerated when they receive the study drug for the first time (according to CTCAE 5.0, the infusion-related reaction is ≤ grade 1), the follow-up infusion time can be 60~90 min (which can be adjusted according to the actual situation).Taxanes is used according to the instructions.
  Arms: Cohort 4
Biological: IAE0972+Capecitabine — IAE0972: every 21 days is defined as a treatment cycle, and IAE0972 is infused intravenously on the 1d, 8d and 15d of each cycle. The first infusion time is about 120 min (which can be adjusted according to the actual situation); If the subjects are well tolerated when they receive the study drug for the first time (according to CTCAE 5.0, the infusion-related reaction is ≤ grade 1), the follow-up infusion time can be 60~90 min (which can be adjusted according to the actual situation).Capecitabine is used according to the instructions.
  Arms: Cohort 5

SUMMARY:
Phase II: To evaluate the safety and tolerability of IAE0972 combined with chemotherapy selected by doctors for R/M HNSCC/NPC after failure or progress of ≤2-line system therapy, and to determine the MTD of combined therapy.

Phase III: According to the RECIST 1.1, the effectiveness of IAE0972 combined with chemotherapy regimen chosen by doctors compared with placebo plus chemotherapy regimen chosen by doctors was evaluated through OS in patients with R/M NPC who failed or progressed after treatment with ≤2-line system.

DETAILED DESCRIPTION:
The Phase II is the dose escalation study of IAE0972 combined with the chemotherapy chosen by doctors, aiming at evaluating the safety, tolerance and preliminary effectiveness for patients with R/M HNSCC/NPC;Phase III aims to evaluate the effectiveness and safety of IAE0972+ doctors' chemotherapy compared with doctors' chemotherapy in patients with R/M NPC who have failed or progressed after treatment with ≤2-line system through OS.In the study, the adverse events and reactions were evaluated by clinical observation, vital signs monitoring and laboratory examination, and related samples such as PK and ADA were collected. Taking RECIST 1.1 as the tumor evaluation standard, after the first infusion of the study drug, every two cycles (±7 days, before the next cycle of administration, and the day of administration in this cycle is defined as D1 of the current cycle), the subjects were evaluated for tumor until the disease progressed, new anti-tumor treatment was started, the researchers judged that it was not suitable to continue to participate (such as intolerable adverse reactions), lost the visit, and voluntarily withdrew.When the subject withdraws from or terminates the treatment (+7 days), the subject should be visited before starting the new anti-tumor treatment (except death and lost visit), and relevant laboratory tests and ADA sample collection should be carried out; After that, their OS was followed up by telephone every 12 weeks (±7 days) until they were lost or died.

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18~75 years old (including the critical value), regardless of gender.
2. Phase II cohort 1, cohort 2: locally advanced squamous cell carcinoma of the head and neck which only occurred in the oral cavity, oropharynx, hypopharynx and larynx after histological diagnosis or had no indication of radical local treatment; In the past, I only received ≤2 line therapy for recurrent and metastatic head and neck squamous cell carcinoma.
3. Phase II cohort 3, cohort 4, cohort 5: Histologically confirmed nasopharyngeal carcinoma, stage IVb or recurrent nasopharyngeal carcinoma that is not suitable for local treatment according to the TNM of AJCC nasopharyngeal carcinoma in the 8th edition of 2017; In the past, they only received ≤2 line therapy for recurrent and metastatic nasopharyngeal carcinoma.
4. According to the researcher's judgment, the chemotherapy in this experiment is applicable.
5. According to the RECIST 1.1 standard, there is at least one measurable lesion (tumor lesions located in previous radiotherapy areas or other local regional treatment sites are generally not regarded as measurable lesions, unless the lesions make clear progress or persist after radiotherapy for three months).
6. The score of physical condition of the ECOG is 0~1.
7. The estimated survival time is ≥3 months.
8. Have sufficient organ functions:

   * Blood system (no blood transfusion or hematopoietic stimulating factor treatment within 14 days): ANC≥1.5×109/L, PLT≥90×109/L, HGB≥ 90 g/L; ② Liver function: TBIL≤1.5 times the ULN, except Gilbert syndrome; AST and ALT are ≤3.0 times ULN, while subjects with liver metastasis or liver cancer need AST and ALT≤3.0 times ULN and total bilirubin ≤ 3.0 times ULN;

     * Renal function: Cr≤1.5 times ULN; If the creatinine is more than 1.5 times ULN, the CCR should be ≥ 50 ml/min (calculated according to Cockcroft-Gault formula);

       * Coagulation function: INR≤1.5 times ULN, APTT≤1.5 times ULN, and INR and APTT≤2.5 times ULN for patients with liver metastasis or liver cancer.
9. Qualified fertile subjects (male and female) must agree to use reliable contraceptive methods (hormone or barrier method or abstinence) with their partners during the trial and at least 6 months after the last medication; The blood pregnancy test of female subjects of childbearing age must be negative within 7 days before the first use of the study drug.
10. Subjects must give informed consent to this study before the experiment, and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Having received chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks before the first use of the investigating drug, the following drugs should be excluded according to the following criteria:

   ① Nitrosourea or mitomycin C was used within 6 weeks before the first use of the study drug;

   ② Oral administration of fluorouracil and small molecule targeted drugs 2 weeks before the first use of the study drug or within 5 half-lives of the drug (whichever is longer);

   ③ Chinese patent drugs with anti-tumor indications were used within 2 weeks before the first use of the study drugs.
2. Received other unlisted clinical research drugs or treatments within 4 weeks before using the research drugs.
3. The adverse reactions of previous anti-tumor treatments have not recovered to NCI CTCAE 5.0 grade evaluation ≤1 grade or the relevant provisions of the selection criteria (except for the toxicity that the researchers judged to have no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, hypothyroidism stabilized by hormone replacement therapy, etc.).
4. It is known that it has hypersensitivity to any antibody drugs (NCI CTCAE 5.0 rating is ≥3), or it has hypersensitivity to research drugs, active ingredients or inactive excipients of chemotherapy schemes.
5. Have received major surgery (excluding puncture biopsy), major trauma or need to undergo elective surgery during the trial within 4 weeks before the first use of the study drug.
6. Having received systemic corticosteroids (prednisone > 10 mg/day or similar drugs with the same dose) within 14 days before the first use of the study drug, except for the following cases: using topical, ophthalmic, intra-articular and intranasal corticosteroids; Short-term use of glucocorticoids for preventive treatment (for example, prevention of contrast agent allergy).
7. Treatment with other immunosuppressants within 28 days or 5 half-lives (whichever is longer) before the first use of the study drug.
8. Have used immunomodulatory drugs within 14 days before the first use of the study drug (Appendix 5).
9. Have been vaccinated with any live vaccine within 4 weeks before the first use of the study drug.
10. Received allogeneic hematopoietic stem cell transplantation or organ transplantation in the past.
11. Brain parenchymal metastasis or meningeal metastasis with clinical symptoms.
12. It has active infection and needs intravenous anti-infection treatment at present.
13. Have a history of immunodeficiency disease, including positive detection of HIV antibody.
14. Active hepatitis B (HBsAg positive and HBV-DNA positive or above the upper limit of normal value) and active hepatitis C (HCV antibody positive and HCV RNA positive or above the upper limit of normal value).
15. Having serious and uncontrollable lung diseases (severe infectious pneumonia, interstitial lung disease, etc.).
16. Have a serious history of cardiovascular and cerebrovascular diseases, including but not limited to:

    ① Severe cardiac rhythm or conduction abnormality, such as ventricular arrhythmia requiring clinical intervention and II-III degree atrioventricular block;

    ② The mean QT interval (QTcF) corrected by Fridericia method was≥470 ms；

    ③ Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events of grade 3 or above occurred within 6 months before the first administration; (4) There is heart failure or LVEF less than 50% with the NYHA cardiac function classification ≥II or structural heart disease with high risk judged by other researchers;

    ⑤ Clinically uncontrollable hypertension.
17. Suffering from active autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), with the exception of clinically stable autoimmune thyroiditis, type I diabetes, vitiligo, cured atopic dermatitis in children, psoriasis that does not require systemic treatment (within the past 2 years), etc.
18. Suffering from other malignant tumors within 5 years before the start of study administration, except for the following cases: malignant tumors that can be expected to be cured after treatment (including but not limited to thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer or breast ductal carcinoma in situ treated by radical surgery).
19. There is clinically uncontrollable effusion in the third space, which is judged by the researcher to be unsuitable for the group.
20. Known alcohol or drug dependence.
21. Have mental disorder or poor compliance.
22. Pregnant or lactating women.
23. The researcher thinks that the subject has other serious history of systemic diseases, or is not suitable to participate in this clinical study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by CTCAE v5.0. | up to 2 years
  AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE is presented.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2 years
  OS is defined as the time from the date of first dosing to death from any cause
Objective response rate (ORR) | up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1
Disease control rate (DCR) | up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1
Progression-free survival (PFS) | up to 2 years
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1 criteria) or death from any cause (whichever occurs first)

IPD SHARING:
Plan to Share IPD: No